CLINICAL TRIAL: NCT05746702
Title: Kronik Obstrüktif Akciğer Hastalığında Yürüyüş Sırasında Yürüyüşün Zaman Mesafe Karakteristikleri ve Kol Salınımlarının İncelenmesi
Brief Title: Investigation of Arm Swings Characteristics in Patient With Chronic Obstructive Pulmonary Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO 22/903
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Chronic Obstructive Pulmonary Disease; Postural; Defect; Gait, Unsteady; Dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Gait Disorders, Neurologic; Dyspnea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The former aim of this study is to determine whether the arm swings change in patients with Chronic Obstructive Pulmonary Disease (COPD) according to healthy subjects. The latter purposes to investigate the correlation between balance parameters and arm swing, how to change arm swing according to severity of the disease, and to determine the relationship between balance and the severity of disease, the relationship of posture both arm swing and severity of disease in patients with COPD. In accordance with this purposes, 20 patients with COPD who have Global Initiative for Chronic Obstruction Lung Disease (GOLD) stage 1-2-3 and 20 healthy controls will be included between the ages of 40 and 65, respectively. Tests and questionnaires will be used in order to determine the severity of COPD and to evaluate posture. Berg Balance Scale, Time Up and Go Test, 6 Minute Pegboard and Ring Test, 6 Minute Walk Test and gait analysis will be performed. It is expected that by determining the parameters that can be affected by severity of COPD. It is estimate to have information about severity of the disease by means of observational analysis. It will guide professional working in the field.

ELIGIBILITY:
Inclusion Criteria:

* Who has been clinically stable for the last 4 weeks,
* who will be able to walk independently for 6 minutes,
* According to the Classification of Airflow Limitation in COPD (GOLD) system, the Stage is 1-2-3,
* who declares that he has not taken part in any other research

Exclusion Criteria:

* walking assistive devices,
* receiving chronic oxygen therapy,
* with central and peripheral vestibular disease,
* with orthopedic, neuromuscular, neurological and cardiac diseases that may affect gait and balance,
* with a history of lung cancer, sarcoidosis, tuberculosis and/or lung surgery,
* who has communication problems,
* with mental and cognitive problems

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred by the department of chest diseases of Hacettepe university will be taken.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-19 (Estimated); Study Completion 2024-10-19 (Estimated)

PRIMARY OUTCOMES:
Arm Swings Characteristics | 1 day
  Change of the arm swings during 6 minute gait in patients with Chronic Obstructive Pulmonary Disease according to healthy subjects.

SECONDARY OUTCOMES:
Spatiotemporal Characteristic | 1 day
  Change of the spatiotemporal characteristic during 6 minute gait in patients with Chronic Obstructive Pulmonary Disease according to healthy subjects.
Upper Extremity Functional Capacity | 1 day
  Upper extremity functional capacity by 6 minute pegboard and ring test in patient with Chronic Obstructive Pulmonary Disease
Balance | 1 day
  Balance by Berg Balance Scale and Time Up Go Test in patient with Chronic Obstructive Pulmonary Disease
Severity of Disease | 1 day
  severity of disease by GOLD ( Global İnitiative for Chronic Obstructive Pulmonary Disease) , CAT ( Chronic Respiratory Questionnaire), Pulmonary Function Test in patient with Chronic Obstructive Pulmonary Disease
Posture | 1 day
  posture by Corbin Posture Analyses Form in patient with Chronic Obstructive Pulmonary Disease
Functional Exercise Capacity | 1 day
  Functional exercise capacity by six minute gait test in patients with Chronic Obstructive Pulmonary Disease.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Demirel, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Aynur Demirel, Ankara, Turkey (Türkiye)